CLINICAL TRIAL: NCT00003149
Title: Phase II of Interleukin-12 for Plateau Phase Multiple Myeloma
Brief Title: Interleukin-12 in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065934; E-1A96
Record Dates: First submitted 1999-11-01; First posted 2004-03-30 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2009-03

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Interleukin-12 Subunit p35

INTERVENTIONS:
Biological: recombinant interleukin-12

SUMMARY:
RATIONALE: Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person's blood cells to kill multiple myeloma cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of interleukin-12 given at different times in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the antitumor activity of interleukin-12 (IL-12) in patients with plateau phase multiple myeloma. II. Evaluate the toxic effects of IL-12 in these patients. III. Evaluate the effectiveness of IL-12 in augmenting T helper subsets in these patients.

OUTLINE: This is a randomized study. Patients are stratified by prior bone marrow transplantation (yes vs no) and by prior pneumococcal vaccine (Pnu-Immune-23) (yes vs no or unknown). Patients are randomized to one of two treatment arms: Arm I: Patients receive Haemophilus influenzae b vaccine (Hib TITER) and Pnu-Immune-23 on day 1 during week 1. Patients who have received Pnu-Immune-23 within the past 3 years receive Hib TITER but no Pnu-Immune-23. Patients receive low dose interleukin-12 (IL-12) subcutaneously (SQ) twice a week during weeks 1 and 2. Beginning on day 1 of week 3, patients receive high dose IL-12 SQ twice a week for an additional 12 weeks. Arm II: Patients receive Hib TITER and Pnu-Immune-23 as in arm I. Patients undergo observation during weeks 1-4, then receive low dose IL-12 SQ twice a week during weeks 5 and 6. Beginning on day 1 of week 7, patients receive high dose IL-12 SQ twice a week for an additional 12 weeks. Both arms: Patients without disease progression may continue to receive high dose IL-12 for an additional 14 weeks. Patients are followed every 3 months for the first 2 years, every 6 months for the next 3 years, and then annually thereafter until death.

PROJECTED ACCRUAL: A total of 40 patients (20 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven plateau phase multiple myeloma at original diagnosis: Bone marrow plasmacytosis with greater than 10% plasma cells, sheets of plasma cells, or biopsy proven plasmacytoma Must be in stable plateau phase requiring objective response, no evidence of continuing improvement by any criteria, and less than 20% variation in M protein at least 4 weeks prior to study Must have at least one of the following at original diagnosis: M protein in serum or urine X-ray evidence of osteolytic lesion Measurable or evaluable M protein Serum M protein greater than 1.0 g/dL Urine M protein greater than 200 mg/24 hours M protein less than these values will be considered evaluable (serum less than 1 g/dL or urine less than 200 mg/24 hours) Nonsecretory patients are ineligible

PATIENT CHARACTERISTICS: Age: 18 and over Performance Status: ECOG 0-2 Life Expectancy: Not specified Hematopoietic: WBC at least 2,500/mm3 Absolute neutrophil count at least 1,250/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) SGOT less than 1.5 times ULN Renal: Creatinine clearance at least 50 mL/min Cardiovascular: No New York Heart Association class III or IV congestive heart failure Other: Not pregnant or nursing Fertile patients must use effective contraception No uncontrolled peptic ulcer disease No inflammatory bowel disease No history of significant autoimmune disease (rheumatoid arthritis or systemic lupus erythematosus)

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 60 days since prior biologic response modifiers At least 60 days since prior bone marrow transplantation Chemotherapy: At least 60 days since prior chemotherapy Endocrine therapy: No concurrent corticosteroids Radiotherapy: Not specified Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1997-12; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Q. Lacy, MD, Study Chair — Mayo Clinic
Locations (10):
- United States (10):
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Ochsner, New Orleans, Louisiana
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of Rochester Cancer Center, Rochester, New York
  - Hahnemann University Hospital, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Lacy MQ, Jacobus S, Blood EA, Kay NE, Rajkumar SV, Greipp PR. Phase II study of interleukin-12 for treatment of plateau phase multiple myeloma (E1A96): a trial of the Eastern Cooperative Oncology Group. Leuk Res. 2009 Nov;33(11):1485-9. doi: 10.1016/j.leukres.2009.01.020. Epub 2009 Feb 24. PMID 19243818